CLINICAL TRIAL: NCT00252239
Title: Phase 2B Study of Tenecteplase (TNK) in Acute Ischemic Stroke (TNK-S2B)
Brief Title: Study of Tenecteplase (TNK) in Acute Ischemic Stroke (TNK-S2B)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, E. Clarke Haley, Professor, Department of Neurology, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11231; R01NS045170 (NIH); R01NS037666 (NIH)
Record Dates: First submitted 2005-11-10; First posted 2005-11-11 (Estimated); Results first posted 2015-01-19 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-02

CONDITIONS: Stroke
Keywords: stroke; tenecteplase; TNK; ischemic; tissue plasminogen activator; tPA
MeSH Terms: conditions — Stroke; Ischemia | interventions — Tenecteplase; Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): tenecteplase
  Interventions: Drug: tenecteplase
- 2 (Active Comparator): tissue plasminogen activator, tPA
  Interventions: Drug: tissue plasminogen activator, tPA

INTERVENTIONS:
Drug: tenecteplase — This study will compare 3 different doses of tenecteplase to tPA.
  Other Names: TNK
  Arms: 1
Drug: tissue plasminogen activator, tPA — To date, tissue plasminogen activator (tPA) is the only scientifically-proven and FDA-approved treatment for acute stroke.
  Other Names: tPA
  Arms: 2

SUMMARY:
The purpose of this study is to determine which of 3 different doses of tenecteplase (TNK) is better for treating stroke patients and if TNK offers an advantage over currently available treatment with tissue plasminogen activator (tPA).

DETAILED DESCRIPTION:
Stroke is the third leading cause of death and a leading cause of adult disability in the United States and worldwide. To date, the only scientifically-proven and FDA-approved treatment for acute stroke is the clot-busting drug, tissue plasminogen activator (tPA). A newer clot-busting drug, tenecteplase (TNK), has chemical properties that make it a potentially safer and more effective drug for treating stroke. Preliminary testing of TNK in patients with acute stroke has been encouraging enough to warrant further testing.

This study, TNK-S2B, will compare three different doses of TNK with standard tPA treatment in patients with acute stroke. Patients will be chosen randomly to receive either TNK or tPA. Neither the patient nor his/her doctor will know which medication the patient received until the study is completely finished.

The first part of the study will look at results of treatment in the first 24 hours to select the best dose of TNK to carry forward into a more detailed comparison with standard tPA treatment. After at least 100-150 pairs of the best dose of TNK and tPA patients have been enrolled, entry into the study will pause, and the outcomes at 3 months after stroke will be compared to see if the results of TNK treatment are sufficiently promising as an improvement over standard treatment to justify expanding the study to find a definitive answer.

The study, which will be conducted in at least 8 large medical centers, is expected to last about 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least a serious, measurable deficit on the NIH Stroke Scale in language (aphasia score > 1), motor power (arm or leg > 1), vision (best visual score > 2), or attention (attention score > 2). Thus eligible patients may have a minimum total score of 1 if the deficit is in language or motor power. There is no maximum score that is exclusionary; even patients with severe hemispheric or brainstem deficits will be eligible, as is current practice with intravenous rt-PA. Patients with all ischemic stroke types and in all vascular distributions are eligible.
* Must arrive at participating hospital and treatment begun within 3 hours of the onset of symptoms. Patients awakening with new symptoms must use the time last observed to be normal and awake and the total time cannot exceed three hours prior to treatment as the time of onset.
* Must be 18 years of age or older.

Exclusion Criteria:

* Patients with a) minor stroke symptoms (e.g., sensory loss, ataxia, dysarthria, or facial weakness alone) or b) major symptoms which are rapidly improving by the time of treatment.
* Patients for whom a complete NIH Stroke Score cannot be obtained (e.g., intubated patients or complete amputees).
* Patients with evidence of intracranial hemorrhage on pretreatment CT scan.
* Patients with a clinical presentation that suggests subarachnoid hemorrhage, even if the initial CT scan is normal.
* Patients who are known or suspected to be pregnant.
* Patients with a known bleeding diathesis or patients with a platelet count < 100,000. For patients who are taking oral Warfarin (Coumadin), the results of the pretreatment International Normalized Ratio (INR) must be available prior to treatment and must be
* </= 1.4. Patients who have received heparin within 48 hours must have a normal partial thromboplastin time (PTT) to be eligible. Patients who have received low molecular weight heparin or heparinoid within 24 hours are also excluded.
* Patients with major surgery or serious trauma excluding head trauma within 14 days or serious head trauma within 3 months.
* Patients with a history of gastrointestinal or urinary tract hemorrhage in the previous 21 days.
* Patients with an arterial puncture at a non-compressible site or a lumbar puncture in the previous 7 days.
* Patients who, on repeated measurement, have a systolic blood pressure > 185, or a diastolic blood pressure > 110 mmHg when treatment is to begin, or require aggressive treatment to reduce blood pressure to within these limits.
* Patients with a history of stroke in the previous 3 months or have ever had an intracranial hemorrhage considered to put them at increased risk for intracranial hemorrhage.
* Patients with a serious medical illness likely to interfere with treatment or treatment might adversely affect that illness.
* Patients with abnormal blood glucose thought to account for the neurological deficit.
* Patients with a clinical presentation consistent with acute myocardial infarction or patients with presentation suggesting post-myocardial infarction pericarditis.
* Patients with a seizure at onset of stroke thought to be presenting with post-ictal paralysis mimicking stroke.
* Patients with pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations.
* Patients who have received any other investigational drug within 14 days.
* Patients who have large areas (greater than one lobe) of obvious low density on the baseline CT scan will be presumed to have had ongoing cerebral ischemia for greater than 3 hours, and will, therefore, be excluded. Patients with subtle early signs of cerebral infarction (e.g., sulcal effacement, blurring of the grey-white junction, asymmetry of the basal ganglia, insular ribbon sign, and others) and the dense artery sign on baseline CT scan will be eligible. Similarly, evidence of previous remote cerebral infarction on baseline CT will not be exclusionary.
* Patients for whom informed consent cannot be obtained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2005-11; Primary Completion 2009-03 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Clarke Haley, Jr., M.D., Principal Investigator — Clinical Coordinating Center, Department of Neurology, University of Virginia Health System; John L. P. Thompson, Ph.D., Principal Investigator — Statistical Analysis Center, Department of Biostatistics, Mailman School of Public Health
Locations (9):
- United States (9):
  - University of California at San Diego, San Diego, California
  - Colorado Neurological Institutes, Englewood, Colorado
  - Johns Hopkins-Bayview Medical Center, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Long Island Jewish Hospital, New Hyde Park, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University, Statistical Analysis Center, New York, New York
  - University of Texas at Houston, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia

REFERENCES:
- [Derived] Haley EC Jr, Thompson JL, Grotta JC, Lyden PD, Hemmen TG, Brown DL, Fanale C, Libman R, Kwiatkowski TG, Llinas RH, Levine SR, Johnston KC, Buchsbaum R, Levy G, Levin B; Tenecteplase in Stroke Investigators. Phase IIB/III trial of tenecteplase in acute ischemic stroke: results of a prematurely terminated randomized clinical trial. Stroke. 2010 Apr;41(4):707-11. doi: 10.1161/STROKEAHA.109.572040. Epub 2010 Feb 25. PMID 20185783

RESULTS

PARTICIPANT FLOW:
Groups:
- TNK 0.1 mg/kg: Lowest dose tenecteplase
- TNK 0.25 mg/kg: Medium dose tenecteplase
- TNK 0.4 mg/kg: Highest dose tenecteplase
- tPA 0.9 mg/kg: tissue plasminogen activator, tPA
  tissue plasminogen activator, tPA: To date, tissue plasminogen activator (tPA) is the only scientifically-proven and FDA-approved treatment for acute stroke.
Period: Overall Study
Arm/Group | TNK 0.1 mg/kg | TNK 0.25 mg/kg | TNK 0.4 mg/kg | tPA 0.9 mg/kg
Started | 31 | 31 | 19 | 31
Completed | 30 | 31 | 17 | 30
Not Completed | 1 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TNK 0.1 mg/kg | TNK 0.25 mg/kg | TNK 0.4 mg/kg | tPA 0.9 mg/kg | Total
Number analyzed (Participants) | 31 | 31 | 19 | 31 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (19) | 69 (15) | 68 (16) | 72 (16) | 69 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 15 | 6 | 14 | 54
  Male | 12 | 16 | 13 | 17 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 4 | 4 | 5 | 18
  White | 24 | 26 | 12 | 25 | 87
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 1 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 31 | 31 | 19 | 31 | 112

OUTCOME MEASURES:

1. Primary Outcome: Functional Handicap (Modified Rankin Score)
Description: The scale range is from 0 (perfect health without symptoms) to 6 (death). Percentage of participants with Modified Rankin Score >=4 are reported.
Time Frame: 3 months
Measure: Number; unit: percentage of participants
Arm/Group | TNK 0.1 mg/kg | TNK 0.25 mg/kg | TNK 0.4 mg/kg | tPA 0.9 mg/kg
Number analyzed (Participants) | 31 | 31 | 19 | 30
percentage of participants | 22.6 | 35.5 | 31.6 | 32.3

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | TNK 0.1 mg/kg | TNK 0.25 mg/kg | TNK 0.4 mg/kg | tPA 0.9 mg/kg
Serious Adverse Events (participants affected / at risk) | 13/31 | 25/31 | 13/19 | 26/31
Other Adverse Events (participants affected / at risk) | 25/31 | 24/31 | 17/19 | 20/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TNK 0.1 mg/kg (N=31) | TNK 0.25 mg/kg (N=31) | TNK 0.4 mg/kg (N=19) | tPA 0.9 mg/kg (N=31)
Hemorrhage, CNS (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1) — Symptomatic hemorrhage defined as clinically important neurological worsening lasting more than 8 hours and judged by independent adjucator to have been caused by blood seen on head CT scanning
Hemorrhage/Bleeding - other (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Retroperitoneal hemorrhage
Infection with unknown ANC (General disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Vascular - other (Vascular disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Cardiac General (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Death not associated with CTCAE term (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Elevated creatinine (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Reduced hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection with Grade 3 or 4 neutrophils (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection with normal, Grade 1 or 2 neutrophils (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignancy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal/soft tissue - other (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neurology-other (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sodium, serum high (hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Valvular heart disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel injury - artery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CNS ischemia (Nervous system disorders) | 5 (5) | 7 (7) | 5 (5) | 7 (7)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TNK 0.1 mg/kg (N=31) | TNK 0.25 mg/kg (N=31) | TNK 0.4 mg/kg (N=19) | tPA 0.9 mg/kg (N=31)
Pain (General disorders) | 14 (14) | 8 (8) | 6 (6) | 4 (4)
Blood/Bone marrow - other (Blood and lymphatic system disorders) | 5 (5) | 6 (6) | 5 (5) | 5 (5)
Hemoglobin low (Blood and lymphatic system disorders) | 4 (4) | 9 (9) | 4 (4) | 4 (4)
Potassium, serum low (Metabolism and nutrition disorders) | 5 (5) | 6 (6) | 4 (4) | 3 (3)
Bruising in absence of grade 3 or 4 thrombocytopenia (Skin and subcutaneous tissue disorders) | 2 (2) | 7 (7) | 2 (2) | 5 (5)
Metabolic/laboratory - other (Metabolism and nutrition disorders) | 5 (5) | 3 (3) | 3 (3) | 4 (4)
Constipation (Gastrointestinal disorders) | 3 (3) | 4 (4) | 3 (3) | 1 (1)
Glucose, serum-high (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 4 (4) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 3 (3) | 5 (5)
Nausea (General disorders) | 3 (3) | 3 (3) | 3 (3) | 2 (2)
Calcium, serum low (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 1 (1) | 3 (3)
Hemorrhage, CNS (Nervous system disorders) | 0 (0) | 4 (4) | 4 (4) | 2 (2) — Asymptomatic blood on head CT scan not accompanied by neurological worsening
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 4 (4) | 2 (2) | 2 (2)
Mood alteration (Psychiatric disorders) | 1 (1) | 5 (5) | 2 (2) | 2 (2)
Albumin, serum low (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 1 (1) | 3 (3)
Valvular heart disease (Cardiac disorders) | 2 (2) | 3 (3) | 1 (1) | 3 (3)
Cardiac general - other (Cardiac disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Hemorrhage, GU (Renal and urinary disorders) | 0 (0) | 1 (1) | 4 (4) | 3 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
Fever, in the absence of neutropenia (General disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2)
Hemorrhage, GI (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Magnesium, serum low (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Neutrophils/granulocytes high (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Pancreatic endocrine: glucose intolerance (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
Premature termination limits any conclusions from the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No